CLINICAL TRIAL: NCT04258241
Title: The Efficacy of Local Infiltration Analgesia for Postoperative Pain Management and Functional Recovery After Total Knee Arthroplasty: Peripheral Nerve Blocks With and Without Local Infiltration Analgesia
Brief Title: The Efficacy of Local Infiltration Analgesia for Postoperative Pain Management After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Inna Jaremko, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEC-MF-36
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Primary Total Knee Arthroplasty
Keywords: Local infiltration analgesia; Primary knee arthroplasty; Postoperative pain management; Postoperative recovery; Adductor canal block; Femoral triangle block
MeSH Terms: interventions — Anesthetics, Local; Needles; Solutions; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local infiltration analgesia with local anesthetic (LIA+) (Active Comparator): Local infiltration analgesia will be performed at the end of the surgery by injection of 150 mg of bupivacaine, 0.3 mg of epinephrine and 90 ml of normal saline.
  Interventions: Procedure: Local infiltration analgesia with local anesthetic; Device: Needle; Drug: Solution with local anesthetic
- Local infiltration analgesia without local anesthetic (LIA-) (Placebo Comparator): Local infiltration analgesia will be performed at the end of the surgery by injection of 0.3 mg of epinephrine and 120 ml of normal saline.
  Interventions: Procedure: Local infiltration analgesia without local anesthetic; Device: Needle; Drug: Solution without local anesthetic

INTERVENTIONS:
Procedure: Local infiltration analgesia with local anesthetic — The orthopedic surgeon will perform local infiltration analgesia at the end of the surgery. The knee joint capsule, periarticular and subcutaneous tissues will be infiltrated with 150 mg of bupivacaine, 0.3 mg of epinephrine and 90 ml of normal saline.
  Arms: Local infiltration analgesia with local anesthetic (LIA+)
Procedure: Local infiltration analgesia without local anesthetic — The orthopedic surgeon will perform local infiltration analgesia at the end of the surgery. The knee joint capsule, periarticular and subcutaneous tissues will be infiltrated with 0.3 mg of epinephrine and 120 ml of normal saline.
  Arms: Local infiltration analgesia without local anesthetic (LIA-)
Device: Needle — 18-gauge 40 mm Sterican needle (B. Braun Medical Inc., Melsungen, Germany) will be used to perform local infiltration analgesia.
Drug: Solution with local anesthetic — Solution of 150 mg of bupivacaine, 0.3 mg of epinephrine and 90 ml of normal saline will be used to perform local infiltration analgesia.
  Other Names: Containing bupivacaine
  Arms: Local infiltration analgesia with local anesthetic (LIA+)
Drug: Solution without local anesthetic — Solution of 0.3 mg of epinephrine and 120 ml of normal saline will be used to perform local infiltration analgesia.
  Other Names: Without bupivacaine
  Arms: Local infiltration analgesia without local anesthetic (LIA-)

SUMMARY:
This prospective, double-blinded, randomized controlled study evaluates the effects of peripheral nerve blocks with and without local infiltration analgesia for postoperative pain management after primary total knee arthroplasty. There are no any studies that show the demand for local infiltration analgesia when together peripheral nerve blocks are performed. Patients undergoing primary total knee arthroplasty will be randomly assigned to receive local infiltration analgesia with or without (placebo group) local anesthetic. All patients will receive peripheral nerve blocks for postoperative analgesia: femoral triangle and distal adductor canal blocks. Comparison of these two groups of patients will be based on the effects on postoperative pain control, the extent of motor blockade, the ability of early leg motion and ambulation, patients satisfaction rates over the time of clinical recovery.

Consequently, the investigators hypothesized that peripheral nerve blocks (femoral triangle and distal adductor canal blocks) with and without local infiltration analgesia provide similar postoperative pain relieving effects and the ability of early mobilization after total knee arthroplasty.

DETAILED DESCRIPTION:
The aim: to evaluate peripheral nerve blocks with and without local infiltration analgesia regarding the postoperative analgesic efficacy, the ability of early motion and ambulation in patients following primary total knee arthroplasty.

Primary Hypothesis: peripheral nerve blocks with (LIA+) and without (LIA-) local infiltration analgesia provide similar postoperative pain relieving effects after primary total knee arthroplasty.

Secondary Effects: peripheral nerve blocks with (LIA+) and without (LIA-) local infiltration analgesia provide similar ability to recover after primary total knee arthroplasty.

The objectives:

1. To compare postoperative pain control effects between LIA+ and LIA- groups of patients after primary total knee joint replacement surgery.
2. To assess the ability of early motion and ambulation after total knee joint replacement surgery between the LIA+ and LIA- groups.
3. To estimate opioid consumption and its adverse effects in LIA+ and LIA- groups of patients after primary total knee arthroplasty.
4. To compare the patient's postoperative satisfaction rates in LIA+ and LIA- groups of patients after primary total knee arthroplasty.

Methods:

The prospective, double-blinded study includes American Society of Anesthesiologists (ASA) I-III patients, aged 18-90 years, admitted for primary total knee arthroplasty. Preoperatively patients will be blindly randomized into one of two groups: LIA+ (peripheral nerve blocks with local infiltration analgesia) and LIA- (placebo group, peripheral nerve blocks without local infiltration analgesia). Group assignment will be concealed by opaque envelopes that will be opened only after enrollment. The anesthesiologist performing the block will be aware of the treatment, but the participant and outcomes assessor will be blinded to group assignment.

The anesthesiologist will perform peripheral nerve blocks under the guidance of a linear ultrasound transducer probe. The femoral triangle and distal adductor canal blocks will be performed. The femoral triangle block will be performed at the level where the medial border of the sartorius muscle intersects the medial border of the adductor longus muscle with an injection of 10 ml of 0.125% bupivacaine. A local anesthetic will be injected laterally to the femoral artery. The distal adductor canal block will be performed at the level where the femoral vessels (artery and vein) dive deeper from the sartorius muscle with an injection of 10 ml of 0.125% bupivacaine. A local anesthetic will be injected under the femoral artery. The orthopedic surgeon will perform local infiltration analgesia with 150 mg of bupivacaine, 0.3 mg of epinephrine and 90 ml of normal saline in LIA+ group and with 0.3 mg of epinephrine together with 120 ml of normal saline in LIA- group.

At the perioperative period, all patients from both groups will receive a standardized anesthetic and analgesic. Premedication of midazolam 2.5-5 mg and dexamethasone 4 mg will be given to all patients and a slow fluid infusion of crystalloids with 1 g of tranexamic acid and 10 mg of ketamine started once an intravenous cannula will be placed. Spinal anesthesia after identification of the subarachnoid space will be performed with 15 mg of levobupivacaine. After that, peripheral nerve blocks will be performed under the ultrasound guidance. Patients will be sedated with intravenously administered propofol during the surgery. At the end of the operation, local infiltration with or without bupivacaine (depending on the group of patients) will be performed. After the surgery, patients will be transferred to the post-anesthesia care unit (PACU).

At the postoperative period for analgesia NSAIDs will be available to both groups of patients. NSAIDs such as dexketoprofen 50 mg, acetaminophen 1 g - 3 times per day and dexketoprofen/tramadol 25/75 mg will be administered after the surgery. Opioids will also be available to patients as intramuscular boluses of pethidine 50 mg or morphine 10 mg without restriction and administered for moderate or severe pain (VAS pain score of 5 or greater out of 10).

The postoperative pain control efficacy will be assessed at 3, 6, 24 and 48 hours after the surgery using the visual analogue scale (VAS) from 0 to 10 (0 - no pain, 10 - worst imaginable pain) at rest, during active and passive 45-degree knee flexion. All the requirements of additional analgesics and their adverse effects will be recorded.

The extent of motor blockade and the ability of early motion will be evaluated at 3, 6, 24, 48 hours after the surgery. Patients will be asked to flex the foot, flex the knee and to lift the straight leg. The possible motion at 3, 6, 24 and 48 hours postoperatively will be assessed with the Bromage scale grades: Grade I - free movement of legs and feet; Grade II - just able to flex knees with free movement of feet; Grade III - unable to flex knees, but with free movement of feet; Grade IV - unable to move legs or feet.

The patients ability of early ambulation will be evaluated using the Timed Up and Go (TUG) test at 24 and 48 hours after the surgery. To do the TUG test, patients will have to sit down on the bed, get up from the bed, walk 3 meters forward, turn, walk back 3 meters to the bed and sit down. The time taken by a patient to perform this test will be calculated with a chronometer.

After the conversation with each patient and assessment of the postoperative pain control efficacy, the ability of early postoperative motion and ambulation, the rate of patient satisfaction will be evaluated using a 10 point scale from 0 (completely unsatisfied) to 10 (totally satisfied) at 3, 6, 24, 48 hours after the surgery.

According to the study protocol, both groups of patients will be compared in terms of postoperative pain control, opioid consumption, early motion and ambulation ability, the incidence of complications (if any), and patients satisfaction rates over time of clinical recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total knee arthroplasty under spinal anaesthesia;
* Age 18 - 90 years;
* Patients conformed to American Society of Anaesthesiologists (ASA) physical status I-III in preoperative assessment;
* Ability to follow the study protocol.

Exclusion Criteria:

* Inability or refusal to follow the study protocol.
* American Society of Anesthesiologists (ASA) physical status classification of IV or higher.
* Coagulopathy.
* Pre-exiting lower extremity neuromuscular disorders.
* Local infection over injection site.
* Allergy or contraindications to the drugs used in the study (local anesthetics, NSAIDs, opioids).
* Chronic opioid use.
* Other type of anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Changes in postoperative pain intensity and pain control: VAS pain scale | First 48 hours after primary total knee arthroplasty.
  Postoperative pain will be assessed in both groups using the visual analogue scale (VAS). The VAS pain scale (numerical rating scale) consists of a range from 0 (no pain) to 10 (worst imaginable pain). Higher score indicate greater pain intensity. Interpretation: 0 (no pain); 1-3 (mild pain); 4-6 (moderate pain); 7-10 (severe pain). Pain control will be assessed at rest, during active and passive 45 degree knee flexion at 3, 6, 24, 48 hours after the surgery.

SECONDARY OUTCOMES:
Extent of motor blockade. | First 48 hours after primary total knee arthroplasty.
  The extent of postoperative motor blockade and the ability of early motion will be evaluated using the Bromage scale: Grade I - free movement of legs and feet; Grade II - just able to flex knees with free movement of feet; Grade III - unable to flex knees, but with free movement of feet; Grade IV - unable to move legs or feet. It will be assessed at 3, 6, 24, 48 hours after the surgery.
Postoperative ability of early ambulation. | First 48 hours after primary total knee arthroplasty.
  The postoperative ability of early ambulation will be assessed using the Timed Up and Go (TUG) test. The TUG test measures the time it takes the patient to get up from a bed, walk 3 m, turn, walk back to the bed and sit down. The TUG test results will be evaluated at 24 and 48 hours after the surgery.
Opioid consumption. | First 48 hours after primary total knee arthroplasty.
  The need of additional opioid consumption will be recorded at 3, 6, 24 and 48 hours after the surgery in both groups.
Rate of patients satisfaction: 10 point scale | First 48 hours after primary total knee arthroplasty.
  Patients satisfaction rates will be evaluated using a 10 point scale from 0 (completely unsatisfied) to 10 (totally satisfied) at 3, 6, 24, 48 hours after the surgery.
Number of participants with postoperative complications. | First 48 hours after primary total knee arthroplasty.
  The total number of postoperative complications (medication toxicity, falls) will be counted in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Arunas Gelmanas, MDPhDAssProf, Study Chair — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences Kauno Klinikos, Department of Anesthesiology, Kaunas, Lithuania

REFERENCES:
- [Background] Mont MA, Beaver WB, Dysart SH, Barrington JW, Del Gaizo DJ. Local Infiltration Analgesia With Liposomal Bupivacaine Improves Pain Scores and Reduces Opioid Use After Total Knee Arthroplasty: Results of a Randomized Controlled Trial. J Arthroplasty. 2018 Jan;33(1):90-96. doi: 10.1016/j.arth.2017.07.024. Epub 2017 Jul 25. PMID 28802777
- [Background] Andersen LO, Kehlet H. Analgesic efficacy of local infiltration analgesia in hip and knee arthroplasty: a systematic review. Br J Anaesth. 2014 Sep;113(3):360-74. doi: 10.1093/bja/aeu155. Epub 2014 Jun 17. PMID 24939863
- [Background] Beswick AD, Dennis J, Gooberman-Hill R, Blom AW, Wylde V. Are perioperative interventions effective in preventing chronic pain after primary total knee replacement? A systematic review. BMJ Open. 2019 Sep 6;9(9):e028093. doi: 10.1136/bmjopen-2018-028093. PMID 31494601
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. The Optimal Analgesic Block for Total Knee Arthroplasty. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):711-719. doi: 10.1097/AAP.0000000000000485. PMID 27685346